CLINICAL TRIAL: NCT06669923
Title: Sugar-Sweetened Beverage (SSB) and Racial Disparities of Right Vs Left Colon Epigenetic Aging
Brief Title: Understanding Sugar-Sweetened Beverages (SSB) and Colorectal Cancer (CRC)
Acronym: SSB and CRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Li Li, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSR230101
Record Dates: First submitted 2024-01-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Education as Topic; National Program of Cancer Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baseline (No Intervention): Baseline study collects baseline data and screens for potential participants for the follow-up study.
- Follow Up - Patient Education Group (Sham Comparator)
  Interventions: Behavioral: Patient Education
- Follow Up - iSIPsmarter Program Group (Experimental)
  Interventions: Behavioral: iSIPsmarter Program

INTERVENTIONS:
Behavioral: iSIPsmarter Program — web-based behavioral intervention to reduce sugary drink intake
  Other Names: Sugary Drink Program
  Arms: Follow Up - iSIPsmarter Program Group
Behavioral: Patient Education — website with information about cancer screening and prevention (e.g. screening tests for seven types of cancer)
  Other Names: Cancer Prevention Program
  Arms: Follow Up - Patient Education Group

SUMMARY:
This study will recruit and consent approximately 120 subjects in the baseline study until the follow-up study recruitment goals of 20 subjects is met. This pilot proposal to: Aim 1) assess the feasibility of conducting a randomized controlled trial of iSIPsmarter among high-risk patients with newly detected large colorectal adenoma to reduce Sugar-Sweetened Beverages (SSB) consumption, and Aim 2) examine the investigators' central hypothesis that SSBs contribute to racial disparities in the development of side-specific colon neoplasia via differentially impacting epigenetic aging and methylation of right vs. left normal colon tissues of African-Americans (AA) vs European-Americans (EA). In order to do so, the investigators will first conduct a study to collect baseline information from eligible and interested participants. Behavioral, lifestyle, and genetic information will be collected from participants undergoing a colonoscopy with large polypectomy removal to set up a biobank. The participants enrolled in this study will then be screened for their interest and eligibility in participating in the follow-up study, a randomized iSIPsmarter intervention trial. The investigators will enroll 20 patients in the follow-up study (1:1 ratio intervention vs. control; equal number of AAs and EAs) with newly detected/resected large colorectal adenomas to collect normal colon tissue biopsies pre- and post-iSIPsmarter intervention and test the investigators' hypotheses.

ELIGIBILITY:
Baseline Study:

Inclusion Criteria:

* Patients scheduled for a colonoscopy (large polyp removal)
* Patients 18+

Exclusion Criteria:

* Subjects who do not speak English
* Subjects diagnosed with inflammatory bowel disorder
* Subjects diagnosed with cancer (except non-melanoma skin cancer)
* Subjects taking blood thinners at time of colonoscopy (except 325 mg daily aspirin)

Follow-up Study:

In order to be eligible to participate in the f/up study, an individual must meet all of the criteria for the Baseline study AND:

Inclusion Criteria:

* Regular access (<1/week) to the internet.
* Drink more than recommended amount of sugar-sweetened beverages per day (assessed from participant's responses to the Beverage Questionnaire section (BEVQ-15) of the Computer Administered Phone Interview (CAPI), from the Baseline study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2029-11-15 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sugar-sweetened beverages | Baseline, 9-weeks, 6-months, 18 months
  Measured using the Beverage Questionnaire 15 (BEVQ-15), measured in oz

SECONDARY OUTCOMES:
Degree of physiological aging, assessed by DNA methylation, of right vs. left colorectal tissue biopsies at Baseline and 6 months. | Baseline, 6 months
  Measured by comparing baseline physiological aging of right vs. left colon tissue biopsies with biopsies collected 6 months post-intervention.
Degree of physiological aging, assessed by DNA methylation, of right vs. left colorectal tissue biopsies at Baseline and 18 months. | Baseline, 18 months
  Measured by comparing baseline physiological aging of right vs. left colon tissue biopsies with biopsies collected 18 months post-intervention.
Change from baseline dietary quality as measured by the components of the Healthy Eating Index (HEI) | Baseline, 9-weeks, 6-months, 18 months
  2 unannounced recalls (one weekend and one weekday) using state-of-the-art Nutrition Data System for Research (NDSR) software and multiple pass methods. HEI indicators will be extracted from the NDSR system and examined for changes in the total HEI score, on a 100-point continuous scale (higher scores reflective higher diet quality)

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, PhD, Principal Investigator — UVA, Dept of Family Medicine; Jamie Zoellner, PhD, RD, Principal Investigator — UVA, Dept of Public Health Sciences

IPD SHARING:
Plan to Share IPD: No